CLINICAL TRIAL: NCT04806776
Title: Central Venous Catheter Dressing Change and Bacterial Colonization in Pediatric Intensive Care Unit
Brief Title: Frequence of Dressing Change and Bacterial Colonization in Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xiamen Children's Hospital (Other); Shenzhen Children's Hospital (Other Government); Anhui Province Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FNDGJ202008
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Bacterial Infections
Keywords: Central venous access device; dressing; bacterial colonization; medical adhesive-related skin injury
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24hrs dressing change (Active Comparator): The first dressing change and sampling were completed 24 hours after catheterization in the operating room or PICU Then the second dressing change and sampling were completed 7days later(if there is no clinical indication occur,such leaking,blood).
  Interventions: Other: 24hrs dressings change
- 7d change dressing (Experimental): Dressing change and sampling were completed 7days after catheterization in the operating room or PICU.(if there is no clinical indication occur,such leaking,blood).
  Interventions: Other: 7days dressings change

INTERVENTIONS:
Other: 24hrs dressings change — The first dressing change and sampling were completed 24 hours after catheterization in the operating room or PICU.When bedside nurse remove the dressing ,the researchers used 4 normal saline cotton swabs to wipe the skin under the dressing. Taking the puncture point as the center, 4 cotton swabs wipes 4 points in the northwest, northeast, Southeast and northeast direction 1cm away from the puncture point,separately.Then the specimen delivered to Laboratory..Then the second dressing change and sampling were completed 7days later(if there is no clinical indication occur,such leaking,blood).
  Arms: 24hrs dressing change
Other: 7days dressings change — The first dressing change and sampling were completed 7 days after catheterization in the operating room or PICU.When bedside nurse remove the dressing ,the researchers used 4 normal saline cotton swabs to wipe the skin under the dressing. Taking the puncture point as the center, 4 cotton swabs wipes 4 points in the northwest, northeast, Southeast and northeast direction 1cm away from the puncture point,separately.Then the specimen delivered to Laboratory..(if there is no clinical indication occur,such leaking,blood).
  Arms: 7d change dressing

SUMMARY:
This study is non-inferiority trial design.The relationship between whether dressing change 24hrs after CVC (central venous catheter) catheterization and bacterial colonization of the skin.

DETAILED DESCRIPTION:
Central venous catheter (CVC) was punctured directly through jugular vein, subclavian vein and femoral vein, and its tip is located in superior vena cava or inferior vena cava. CVC is widely used in ICU because of its kinds of advantages. However, CVC, as an invasive puncture method, may bring more complications. The incidence of central line associated bloodstream infection (CLABSI) was 1.33-31.6/1000 catheterization day , and the death rate due to CVC associated bloodstream infection is 3-5% . Therefore, various organizations have formulated guidelines for the prevention of CLABSI and best evidence summary . From October 2019 to April 2020, taking the children's hospital of Fudan University as the leading unit, PICU of children's Hospital Affiliated to Zhejiang University, Anhui children's Hospital, Xiamen children's Hospital, Shenzhen Children's Hospital and Guangzhou Women's and Children's medical center as the cooperation units, carried out children's central venous catheterization Multi center research on best practices of management and maintenance. It was found that changing dressings 24 hours after catheterization may increase the incidence of MARSI, and repeatedly exposing dressings may also increase the incidence of CLABSI. The research team returned to the original evidence and consulted the guidelines. It was found that: under the premise of achieving the maximum aseptic catheterization, the guidelines issued by various institutions did not mention that the application should be replaced 24 hours after catheterization; however, the evidence was mentioned in the evidence summary, but there was no support from the relevant original literature. Therefore, it is worth discussing whether children need to change dressings 24 hours after catheterization. This study is non-inferiority trial design.

ELIGIBILITY:
Inclusion Criteria:

* CVC catheter was placed in the research site (including the operating room and PICU);
* only one CVC catheter was placed during the research time

Exclusion Criteria:

* catheter was inserted from another hospital and in emergency;
* the tip of CVC catheter was not in the upper and lower vena cava;
* children had history of CLABSI before the study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Bacterial colonization in the skin under dressing | 7days or 8days of central venous catheter insertion
  incidence of bacterial colonization in the skin under dressing :7days or 8days after insertion,when nurse change the CVC dressing,The researchers used 4 normal saline cotton swabs to wipe the skin under the dressing. Taking the puncture point as the center, 4 cotton swabs wipes 4 points in the northwest, northeast, Southeast and northeast direction 1cm away from the puncture point,separately. Samples were inoculated on Petri dishes respectively.The type and quantity of bacteria will be reported by the Laboratory. The colony number above 20 CFU(colony-forming units) / cm2 means Bacterial colonization occurred.

SECONDARY OUTCOMES:
Incidence of Medical adhesive-related skin injury(MARSI) | from cvc insertion to 7days or 8days
  MARSI:persistent erythema and / or other skin abnormalities within 30 minutes or more after nurse change the dressings

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gu, doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT04806776/SAP_001.pdf